CLINICAL TRIAL: NCT00946868
Title: Prevalence of Metabolic Syndrome in Patients With Intermittent Claudication
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Nelson Wolosker, PhD, University of Sao Paulo
Other Study IDs: 0143/09
Record Dates: First submitted 2009-07-23; First posted 2009-07-27 (Estimated); Last update posted 2009-07-27 (Estimated); Status verified 2009-07

CONDITIONS: Intermittent Claudication; Metabolic Syndrome X
Keywords: intermittent claudication; metabolic syndrome
MeSH Terms: conditions — Intermittent Claudication; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intermittent claudication patients: Patients with intermittent claudication with metabolic syndrome and patients with intermittent claudication without metabolic syndrome.

SUMMARY:
Metabolic syndrome, a group of cardiovascular risk factors related to insulin resistance, is a major determinant of cardiovascular mortality.

Intermittent claudication is a symptom of an early stage of atherosclerosis.

The aim of this study is to determine the prevalence of the metabolic syndrome in patients with intermittent claudication and its correlation with age, gender, localization of arterial obstruction and association with coronary artery disease.

DETAILED DESCRIPTION:
Studies correlating metabolic syndrome and several illnesses are being published, especially affections associated with atherosclerosis, like coronary artery disease, cerebrovascular disease and peripheral arterial disease.

The term peripheral arterial disease, however, refers to several stages of the development of atherosclerosis in the extremities, comprising since asymptomatic patients as far as individuals with critical ischemia.

Intermittent claudication is a symptom of an early stage of atherosclerosis, when medical interventions may still prevent the progression of the disease. Despite the importance of a precocious diagnosis of metabolic syndrome to initiate adequate treatment, its prevalence among these patients is not well determined in the literature.

This is the biggest casuistic in the literature as far as we know.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with complaints compatible with intermittent claudication of the lower limbs, absence or weakness of arterial pulses on the limb or limbs that are limiting deambulation, ankle-brachial index simila or lower than 0.9

Exclusion Criteria:

* patients with critical limb ischaemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients of the Vascular and Endovascular Department (Intermittent Claudicantion Group)
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2009-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Presence of metabolic syndrome in patients with intermittent claudication | After laboratory exams results.

SECONDARY OUTCOMES:
Correlation of metabolic syndrome with age, sex, localization of the arterial obstruction and the association with symptomatic coronary artery disease. | At the end of data collection

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Wolosker, PhD, Principal Investigator — University of Sao Paulo; Pedro P Leao, PhD, Study Chair — University of Sao Paulo
Locations (1):
- Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Ambrosetti M, Salerno M, Laporta A, Pedretti RF. Metabolic syndrome in patients with intermittent claudication referred to vascular rehabilitation. Int Angiol. 2006 Mar;25(1):14-7. PMID 16520719
- [Result] Ford ES, Giles WH, Mokdad AH. Increasing prevalence of the metabolic syndrome among u.s. Adults. Diabetes Care. 2004 Oct;27(10):2444-9. doi: 10.2337/diacare.27.10.2444. PMID 15451914
- [Result] Ford ES, Giles WH. A comparison of the prevalence of the metabolic syndrome using two proposed definitions. Diabetes Care. 2003 Mar;26(3):575-81. doi: 10.2337/diacare.26.3.575. PMID 12610004
- [Result] Ford ES, Giles WH, Dietz WH. Prevalence of the metabolic syndrome among US adults: findings from the third National Health and Nutrition Examination Survey. JAMA. 2002 Jan 16;287(3):356-9. doi: 10.1001/jama.287.3.356. PMID 11790215
- [Result] Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults. Executive Summary of The Third Report of The National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, And Treatment of High Blood Cholesterol In Adults (Adult Treatment Panel III). JAMA. 2001 May 16;285(19):2486-97. doi: 10.1001/jama.285.19.2486. No abstract available. PMID 11368702
- [Result] National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) final report. Circulation. 2002 Dec 17;106(25):3143-421. No abstract available. PMID 12485966